CLINICAL TRIAL: NCT01991288
Title: Does Saphenous Nerve Block Improve Analgesia After Total Knee Replacement When Used in Combination With Local Infiltration Analgesia? A Prospective Randomised Double Blinded Trial.
Brief Title: Analgesic Efficacy of Saphenous Nerve Block in Total Knee Replacement
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cork University Hospital (Other)
Responsible Party: Principal Investigator, DR. Jassim Rauf, Specialist Registrar, Cork University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: JR-0786-GI
Record Dates: First submitted 2013-11-17; First posted 2013-11-25 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2013-11

CONDITIONS: Post Operative Pain
Keywords: Total Knee Replacement; Bupivacaine; Levobupivacaine; Saphenous Nerve Block; Local Infiltration Analgesia
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine; Levobupivacaine; Epinephrine; Saline Solution

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SNB Saphenous Nerve block (Experimental): Patients received SNB preoperatively at mid thigh level with ultrasound guidance. 10 mls 0.5% bupivacaine was administered for nerve block by the anesthetist. All patients also received peri operative Local Infiltration Analgesia by the surgeon. All patients will receive preoperative oxycontin, peri operative paracetamol and diclofenac. Post operatively all patients received regular paracetamol 1g 6 hourly, Diclofenac sodium 12 hourly and oxycontin 10-20 mg 12 hourly. All patients received standardized spinal block by the same anesthetist, post nerve block for surgery.
  Interventions: Procedure: SNB Saphenous Nerve Block
- NSNB Non Saphenous Nerve Block (Active Comparator): Patients only received Local Infiltration Analgesia. As per protocol all patients received the same pre, peri and post operative analgesia as described in the experimental group. All patients had a standardized spinal block for surgery.
  Interventions: Procedure: NSNB Non Saphenous Nerve Block

INTERVENTIONS:
Procedure: SNB Saphenous Nerve Block — Patients in group SNB received an ultrasound guided SNB (a sub sartorial approach) by a single operator with 10 mls 0.5% bupivacaine. At the end of surgery periarticular knee infiltration of 30 mls 0.5% levobupivacaine + 70 mls 0.9% saline + 0.5 mg adrenaline was performed in a staged fashion by the surgeon, beginning with infiltration of the deep structures on tibial surface at 1mm depth around all exposed tissues, medial and lateral collateral ligament origin, all cut surfaces of extensor mechanism, all cut surface of skin and subcutaneous tissue
  Other Names: Bupivacaine; Levobupivacaine; Adrenaline; 0.9% NaCl
  Arms: SNB Saphenous Nerve block
Procedure: NSNB Non Saphenous Nerve Block — All patients at the end of surgery received periarticular knee infiltration of 30 mls 0.5% levobupivacaine + 70 mls 0.9% saline + 0.5 mg adrenaline, in a staged fashion by the surgeon, beginning with infiltration of the deep structures on tibial surface at 1mm depth around all exposed tissues, medial and lateral collateral ligament origin, all cut surfaces of extensor mechanism, all cut surface of skin and subcutaneous tissue
  Other Names: Levobupivacaine; Adrenaline; 0.9% NaCl
  Arms: NSNB Non Saphenous Nerve Block

SUMMARY:
We hypothesize that preoperative saphenous nerve block (SNB) in combination with periarticular local infiltration provides better post operative pain relief (POPR) profile as compared to local infiltration alone

DETAILED DESCRIPTION:
Introduction:

Local infiltration analgesia (LIA) is considered acceptable after total knee replacements (TKR) in terms of analgesia, ease of performance, early mobilization and early hospital discharge . Continuous femoral nerve block has been used to enhance post op pain relief (POPR) for TKR but at the expense of motor blockade . A Sub sartorial approach to saphenous nerve block (SNB) spares the motor block . To date the role of saphenous nerve block for POPR in TKR has not been evaluated.

Methodology:

In order to test this hypothesis, we proposed to carry out a prospective randomized controlled double blinded (surgeon and assessor) trial study. With institutional ethics approval and having obtained written informed consent from each patient, 20 ASA 1 - 3 patients scheduled to undergo TKR under spinal anesthesia +/- sedation were allocated to one of two groups i.e. Group (SNB): patients receiving SNB sub sartorial approach and Group (NSNB): patients not receiving SNB.

Group allocation was determined using computer generated random number tables. Sealed envelopes were opened on the day of the surgery by the attending anesthetist responsible for the care of the recruited patient.

Postoperative period:

Patients were then assessed for pain at rest and on movement on arrival in recovery and then at 6 , 12 and 24 hrs. Visual analogue scale on a 10 cm straight line was used to assess postoperative pain scores as predictive value of post operative analgesia on rest and movement i.e passive flexion of knee to 30 degree . Patients were assessed for any motor block by using maximum tolerable range of active knee flexion (MKF) and maximum range of straight leg raise(MSLR) on arrival in recovery and at 6, 12 and 24 hrs. All patients received regular paracetamol 1g 6 hourly, diclofenac 75 mg 12 hourly, oxycontin 10-20 mg ( depending on age) 12 hourly and oxynorm 10 mg as rescue analgesia.

ELIGIBILITY:
Inclusion Criteria:

American Society of Anaesthesia (ASA) Grade I-lll patients Undergoing elective Total Knee Arthroplasty Patients able to consent and understand all the components of the study.

Exclusion Criteria:

Demented patients Patients having bilateral Knee Replacements Patients unable to comprehend the use of pain scales Allergy to any of the medications used in the study Renal dysfunction Coagulation disorders Peptic ulcer disease precluding use of non-steroidal anti-inflammatory drugs (NSAIDs) Patients unable to use regular opioid medication Any chronic pain condition other than osteoarthritis of the knee.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-11; Primary Completion 2013-05 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Pain on movement at 24 hours time point post operatively | 24 hours hours time point

SECONDARY OUTCOMES:
pain on movement at 6 and 12 hour time point | 6 and 12 hours time points
pain at rest at 6, 12 and 24 hours time points | 6, 12 and 24 hours time points
Maximum Knee Flexion at 6, 12 and 24 hours time points | 6, 12 and 24 hours time points
Maximum Straight Leg Raise Test at 6, 12 and 24 hours time points | 6, 12 and 24 hours time points
Time to First request for rescue analgesia | 24 hours
Cumulative Opioid consumption in 24 hours | 24 hours
Cumulative opioid consumption till discharge | till discharge time
6 Minute walk test | At 24 hours Post block Conduction

OTHER OUTCOMES:
Time to discharge from hospital | 1 week

CONTACTS AND LOCATIONS:
Overall Officials: George Shorten, FFARCSI, PhD, Study Director — Dept. of Anaesthesia & ICU, Cork University Hospital, Cork, Ireland
Locations (1):
- Dept. of Anaesthesia & Intensive Care Unit, Cork University Hospital, Cork, Cork, Ireland